CLINICAL TRIAL: NCT02779569
Title: Prospective, Open, Multi-center, Double Arm Clinical Trial Evaluating the Efficacy of Ultra Low Dose of Decitabine in Myelodysplastic Syndromes (MDS)
Brief Title: A Clinical Trial Evaluating the Efficacy of Ultra Low Dose of Decitabine in Myelodysplastic Syndromes (MDS)
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: The First Affiliated Hospital with Nanjing Medical University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MDS-ULD-2016; ChiCTR-IPR-16008100 (Other Grant/Funding Number: Chinese Clinical Trial Registry)
Record Dates: First submitted 2016-05-09; First posted 2016-05-20 (Estimated); Last update posted 2017-11-08 (Actual); Status verified 2016-05

CONDITIONS: Myelodysplastic Syndromes (MDS)
MeSH Terms: conditions — Myelodysplastic Syndromes | interventions — Decitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Ultra-low-dose group (Experimental): decitabine was subcutaneously administered at 5 to 7 mg/m2 once daily for successive 3 days at the first week, and once daily at weeks 2 to 4, with a total dose of 60 mg in a 4-week cycle.
  Interventions: Drug: decitabine
- Low-dose group (Active Comparator): decitabine was subcutaneously given at 20 mg/m2 once daily for successive 3 days, with a total dose of 60 mg/m2 in a 4-week cycle.
  Interventions: Drug: decitabine

INTERVENTIONS:
Drug: decitabine

SUMMARY:
To evaluate the safety and clinical efficacy of ultra-low-dose decitabine in Chinese MDS

DETAILED DESCRIPTION:
To develop a highly effective and safe protocol, a multi-center, prospective clinical trial was conducted in China, with aims to evaluate the grade III and IV hematologic toxicity and clinical efficacy of subcutaneous injection of ultra-low-dose decitabine (5 to 7 mg/m2) for treatment of myelodysplastic syndrome (MDS), while decitabine at a dose of 20 mg/m2 as a control.

ELIGIBILITY:
Inclusion Criteria:

1. Men or women aged 18 to 80 years;
2. Patients at high risk of MDS assessed by International Prostate Symptom Score (IPSS);
3. Chronic myelomonocytic leukemia (CMML) patients with abnormal white blood cell counts, extremely low platelet count or organ infiltration (such as hepatomegaly, splenomegaly) that required therapy;
4. Patients at low risk of MDS identified by IPSS score who had secondary MDS, platelet count of < 20*10^9/L, no response to erythropoietin (EPO) (non-5q deletion syndrome) in the presence of disease symptoms or blood transfusion dependence, or no response to EPO/lenalidomide (5q deletion syndrome) in the presence of disease symptoms or blood transfusion dependence;
5. Patients with a Eastern Cooperative Oncology Group (ECOG) of 0 to 2;
6. Patients with an expected lifespan of over 6 months;
7. Patients with a aspartate aminotransferase (AST) of < 2.5 times higher than the normal upper limit, alanine aminotransferase (ALT) of < 2.5 times higher than the normal upper limit, total bilirubin of < 1.5 times higher than the normal upper limit, and serum creatinine of < 1.5 times higher than the normal upper limit;
8. Subjects who had recovery of toxicity, did not undergo any therapy 4 weeks prior to the first trial, and did not receive nitrosourea therapy and bone marrow transplantation 6 weeks prior to the first trial;
9. Female subjects were menopausal, underwent surgical sterilization, or had effective contraception (oral contraceptive, injectable contraceptive, intrauterine device, contraceptive patch, male sterilization) prior to enrollment and during the trial, and were negative for serum or urine pregnancy test at screening;
10. No insemination was given to male subjects during the treatment and within 2 months post-treatment;
11. Subjects complying with the study protocol;
12. Subjects that signed the informed consent, which indicated they understood the purpose, the procedure and potential benefits of the trial and were willing to participate in the trial.

Exclusion Criteria:

1. Patients that were diagnosed as acute myeloid leukemia (primitive bone marrow cell proportion of 20% or higher) or other progressive malignant diseases;
2. Patients that received treatment with other drugs within 30 days prior to the first administration of decitabine;
3. Patients that received radiotherapy within 14 days prior to the first administration of decitabine;
4. Patients with uncontrolled heart disease or congestive heart failure;
5. Patients with uncontrolled restrictive or obstructive pulmonary disease;
6. Patients with active viral, bacterial or invasive fungal infections;
7. Patients that were complicated by autoimmune hemolytic anemia or immune thrombocytopenia;
8. Patients with a history of use of azacitidine or decitabine;
9. Patients that were sero-positive for HIV;
10. Patients with mental or other disorders that cannot completely cooperate with the treatment or follow up;
11. Patients bone marrow cannot be sampled;
12. Subjects that were allergic to decitabine vehicle;
13. Pregnant or lactating women.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2016-03; Primary Completion 2019-03 (Estimated); Study Completion 2019-08 (Estimated)

PRIMARY OUTCOMES:
Grade III and IV hematologic toxicity, according to National Cancer Institute common toxicity criteria (NCI-CTC) V3.0 criteria | 8 months

SECONDARY OUTCOMES:
Complete response, according to International Working Group (IWG) response criteria | 8 months
Complete response (CR) rate of bone marrow, according to IWG response criteria | 8 months
Partial response (PR) rate, according to IWG response criteria | 8 months
Hematologic improvement (HI), according to IWG response criteria | 8 months
Overall response rate, defined as CR＋PR＋HI, according to IWG response criteria | 8 months
Cytogenetic response, according to IWG response criteria | 8 months
times of transfusion requirements | 8 months
  times of transfusion requirements during 8 months after enrollment
times of hospitalization | 8 months
  times of hospitalization during 8 months after enrollment
The quality of life, the quality of life will be assessed by European Organization for Research and Treatment of Cancer Quality of Life Questionnaire C30 (EORTC QLQC30) | 8 months

CONTACTS AND LOCATIONS:
Overall Officials: Guangsheng He, Principal Investigator — The First Affiliated Hospital with Nanjing Medical University
Locations (6):
- China (6):
  - No.303 Hospital of Chinese People's Liberation Army, Nanning, Guangxi
  - Jiangsu Province Hospital, Nanjing, Jiangsu
  - Shengjing Hospital of China Medical Univercity, Shenyang, Liaoning
  - The First Affiliated Hospital of Xi'an Jiaotong University, Xi’an, Shanxi
  - People's Hospital of Xinjiang Uygur Autonomous Region, Ürümqi, Xinjiang
  - Zhejiang Provincial Hospital of TCM, Hangzhou, Zhejiang

IPD SHARING:
Plan to Share IPD: Undecided